CLINICAL TRIAL: NCT03253653
Title: Assessing Toxicity of Waterpipe Tobacco Smoking in Laboratory and Naturalistic Settings
Brief Title: Assessing Toxicity of Waterpipe Tobacco Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Nada Kassem, PI, San Diego State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01DA042471-01 (NIH)
Record Dates: First submitted 2017-08-07; First posted 2017-08-18 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Waterpipe Smoking
Keywords: waterpipe; hookah; NNAL; SPMA; 1-HOP; Furan-BDA-NAL; Carbon monoxide; Pulmonary Function
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Intervention Model Description: The investigators will employ a repeated measures design. A sample of 50 adult male and female exclusive WP smokers and a control sample of 25 male and female non-smokers will be recruited. Over a 3-week study, WP smokers will smoke one WP tobacco head during each of 3 separate WP smoking sessions with a 7-day washout period before each session. Session 1, WP smokers will smoke using 1 quick-light charcoal and room temperature water in the WP jar; Session 2, WP smokers will smoke using 1 quick-light charcoal but adding ice cubes to the water in the WP jar; Session 3, WP smokers will smoke WP tobacco without charcoal using an electric WP head and room temperature water. Physiological effects, carbon monoxide exposure and biomarkers of toxicants and carcinogens related to WP tobacco smoking practices will be compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Waterpipe smoking (Experimental): In a repeated measures design, 50 adult male and female exclusive WP smokers will smoke WP tobacco weekly over a 3-week study period with 3 WP smoking practices.
  Interventions: Device: Differential effects of waterpipe smoking practices on toxicity of waterpipe tobacco smoke
- Control (No Intervention): A total of 25 adult make and female nonsmokers will be recruited as a control.

INTERVENTIONS:
Device: Differential effects of waterpipe smoking practices on toxicity of waterpipe tobacco smoke — In a repeated measures design, 50 adult male and female exclusive WP tobacco smokers will smoke WP tobacco weekly over a 3-week study period with 3 WP smoking practices as follows: 1) using room temperature water in the WP jar, 2) adding ice cubes to the water in the WP jar, and 3) using a charcoal-free electronic WP head to heat the tobacco. Six Spot first morning urine samples will be provided by participants. Two urine samples per each of the 3 smoking sessions. Urine samples will be provided on the day of the WP tobacco smoking session and the following day. Physiological measures will be taken at Baseline during the office visit and before and after each of the 3 WP tobacco smoking sessions.
  Arms: Waterpipe smoking

SUMMARY:
Waterpipe smoking is a tobacco use method in which smoke passes through a partially-filled water jar. Burning charcoal heats the waterpipe tobacco which produces the smoke that the user inhales. Waterpipe smoking was associated with increased risk for coronary heart and pulmonary diseases. This Waterpipe Study will inform the FDA on regulating waterpipe tobacco products and reduce the harm of it use. This study will be conducted at homes of hookah smokers, in natural settings, aimed to determine the effects of waterpipe smoking practices on physiological injury markers and biomarkers of toxicity of waterpipe tobacco smoking. The investigators will employ a repeated measures design. The investigators will recruit a sample of 50 adult male and female exclusive waterpipe smokers and a control sample of 25 male and female non-smokers via intercept interviews from San Diego County, California communities. Waterpipe smokers will smoke one waterpipe tobacco head (10g) of Starbuzz during 3 separate sessions with a 7-day washout period before each session, as follows: Session 1, Smoking waterpipe tobacco using 1 quick-light charcoal and room temperature water in the waterpipe jar, Session 2, Smoking waterpipe tobacco using 1 quick-light charcoal and adding ice cubes to the water in the waterpipe jar, and Session 3, Smoking waterpipe tobacco without charcoal using a charcoal-free electrically heated waterpipe head to heat the tobacco, and room temperature water in the waterpipe jar. The following data will be collected: a) Tobacco Use History, b) 4-week Tobacco Exposure Diary, c) Waterpipe Use Session Form, d) Carbon monoxide (CO) exposure: Micro+ Smokerlyzer® CO monitor will be used for exhaled CO pre and 2 minutes post each smoking session, e) Pulmonary function testing and measuring blood pressure, heart rate and respiratory rate, and f) 6 first morning urine samples: pre and post the 3 sessions to measure urinary cotinine, a metabolite of nicotine, 4-(methylnitrosamino)-1- (3-pyridyl)-1-butanol (NNAL) and NNAL-glucuronides (total NNAL), metabolites of the lung carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), 1-hydroxypyrene (1-HOP), a metabolite of the genotoxic carcinogen pyrene, and S-phenylmercapturic acid (SPMA), a metabolite of the human hematotoxicant and leukemogen benzene. The investigators will explore exposure levels to furan, a liver toxicant and carcinogen, among waterpipe smokers via measuring its urinary metabolite, L-2-(acetylamino)-6-(2,5-dihydro-2-oxo-1H-pyrrol-1-yl)-1-hexanoic acid (Furan-BDA-NAL).

DETAILED DESCRIPTION:
Globally, 1 in 3 adults or 1.2 billion people smoke. The World Health Organization (WHO) estimated that tobacco is responsible for the death of 1 in 10 adults worldwide, about 6 million premature deaths each year. In the United States (U.S.), cigarette smoking is responsible for more than 480,000 deaths per year, including nearly 42,000 deaths resulting from secondhand smoke exposure. Tobacco use is the single leading most preventable cause of disease, disability, and mortality in the U.S. Tobacco research tends to focus on cigarettes; however, the rise in waterpipe (WP) tobacco use globally warrants studying all aspects of its toxicity. In 2005, the WHO called for a better understanding of WP tobacco smoking. In 2007, the American Lung Association labeled WP smoking as an emerging deadly trend. WP tobacco use was associated with increased risk for Chronic obstructive pulmonary disease (COPD), heart diseases, lung cancers, oral and esophageal cancers.

COPD is a major public health problem leading to airflow obstruction. In the U.S., tobacco smoke is a key factor in the development of COPD, which was the third leading cause of death in the U.S. in 2014. WP smoking decreases respiratory quality of life in adults. Studies found that pulmonary function following WP smoking was impaired as measured by forced expiratory volume (FEV1), forced vital capacity (FVC), FEV1/FVC, and Forced Expiratory Flow (FEF25-75%). Studies investigating acute cardiovascular injury markers due to WP smoking showed significant increases in heart rate, and in systolic and diastolic blood pressure.

In 2014, the U.S. Food and Drug Administration (FDA) initiated regulation WP tobacco. The FDA proposed that the manufacturers of WP tobacco disclose to the FDA their products' ingredients and report harmful and potentially harmful constituents (HPHCs). A review study showed that exposures to HPHCs are 10-100 times higher in WP tobacco smoke than in cigarette smoke. To inform the FDA on the regulation of WP tobacco products, and reduce the harm of it use, the investigators propose a Waterpipe Project in a natural setting to determine the differential effects of WP smoking practices on physiological injury markers, and biomarkers of toxicants and carcinogens.

Worldwide, the WP is used in Africa, Asia, China, India, and the Middle East. Adolescents and young adults in the U.S. are experimenting with WP smoking. The 2014 U.S. National College Health Assessment II found that nearly one third of U.S. undergraduate college students (38.2% of men and 31.4% of women), reported ever using WP tobacco, and 11.6% of men and 8.3% of women reported current use (past 30 days). Among high school students, the 2013 U.S. National Youth Tobacco Survey showed that 15.1% of boys and 13.5% of girls reported ever WP use.

The WP (hookah) consists of a head, a body, a hose, and a water jar. The tobacco is placed in the head and covered with a perforated aluminum foil to allow air-flow. Burning charcoal is placed on top of the aluminum foil. Upon deep inhalation via the WP hose, suction forces hot air through the head, heating and combusting the tobacco to produce the smoke that is forced down the WP body, into and out of the water in the airtight jar, and through the hose into the smoker's mouth and respiratory system. Smokers inhale charcoal toxicant emissions in addition to those from the WP tobacco. Charcoal combustion contributes greatly to benzene, carbon monoxide (CO) and carcinogenic yields. CO is a smoke toxicant that reduces the blood's ability to transport oxygen to various organs, including the brain, and can cause dizziness, headache, syncope and nausea.

A charcoal-free electrically heated WP head is commercially available. Users were satisfied with this device because they did not have to deal with charcoal fire hazardous ambers and ashes, in addition to enjoying the feeling of reduced harm. WP smokers normally use room temperature water in the WP jar. However, other liquid media are gaining in popularity. According to anecdotal evidence, "adding ice cubes in the WP jar has an enjoyable cooling effect to the inhaled smoke". Smokers practice adding ice cubes at home, and for an extra charge hookah lounges provide this option for customers. Toxic chemicals in WP tobacco smoke include cotinine, a metabolite of the addictive drug nicotine; 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) and NNAL-glucuronides (total NNAL); metabolites of the lung carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK); 1-hydroxypyrene (1-HOP), a metabolite of the genotoxic carcinogen pyrene; and S-phenylmercapturic acid (SPMA), a metabolite of the human hematotoxicant and leukemogen benzene; and Furan-BDA-NAL, a metabolite of the carcinogen furan.

METHODS. will compare exhaled CO, pulmonary functions, blood pressure, heart rate and respiratory rate, and urinary levels of cotinine, NNAL, SPMA, and 1-HOP in first void WP smoker urine samples the morning of, and the morning after a WP smoking session across 3 smoking practices. The investigators will recruit a sample of 50 adult male and female exclusive WP smokers and a control sample of 25 male and female non-smokers. Participants will be recruited and qualified via random intercept screen interviews from San Diego County, California communities. Over a 3-week study period, WP smokers will smoke one WP tobacco head (10g) of Starbuzz during 3 separate sessions with a 7-day washout period before each session in their home in a natural setting: Week 1-Session 1, WP smokers will smoke using 1 quick-light charcoal and room temperature water in the WP jar, Week 2-Session 2, WP smokers will smoke using 1 quick-light charcoal but adding ice cubes to the water in the WP jar, Week 3-Session 3, WP smokers will smoke WP tobacco without charcoal using the electric WP head and room temperature water. The investigators will collect the following forms: a) Tobacco Use History; b) 3-week Tobacco Use and Exposure Diaries; c) WP Smoking Session Day and Exposure Form; and will measure d) CO exposure: Micro+ Smokerlyzer® CO monitor will be used for exhaled CO two minutes pre and post each smoking session; e) Pulmonary function testing and measuring blood pressure, heart rate and respiratory rate pre and post each smoking session; and f) 6 first morning urine samples: pre and post the 3 sessions to measure urinary cotinine, NNAL, 1-HOP, SPMA, and Furan-BDA-NAL. Efforts will be made to recruit equal samples of males and females. Flexible scheduling for study activities where applicable. Proration of incentives will apply for completed activities.

The 3-Week Study period: comprised of 3 WP smoking sessions with 7-day wash-out periods

WP Smoking Session 1. Day 1 - Office Visit: The Office Visit is expected to take between 60 and 90 minutes where potential participants will be trained on the study activities. Consent will be obtained, study forms will be completed, and study related materials such as forms and urine cups will be provided. Scheduling will be arranged for the 3 WP smoking sessions and corresponding home visits. Saliva Test: Trained by the PI, the research assistants (RAs) will use NicAlert, an accurate and valid commercial semi-quantitative instant saliva cotinine test, to validate non-smoking status, which the investigators used successfully in their previous studies. The following physiological baseline data will be collected: pulmonary functions, blood pressure, heart rate and respiratory rate. Days 2 - 6: The RAs will contact participants by phone on the 4th day to confirm adherence to the 7-wash-out period and diaries, and on the 6th day to remind participants to collect the first morning urine sample on day 7, and to arrange for a home visit for the first WP smoking session. Day 7: WP smoking session 1. WP smokers will provide one first morning urine sample and store it in their refrigerator (freezer section). WP smokers will smoke WP tobacco (10 grams) as they normally do using charcoal and room temperature water in the water jar. The RAs will collect expired CO levels 2 minutes before and 2 minutes after concluding smoking, and will measure pulmonary functions, blood pressure, heart rate and respiratory rate thereafter. Day 8: Participants will provide a first morning urine sample. The RAs will pick up the 2 urine samples (frozen in a cooler to transfer them to the research center laboratory), and arrange for the 2nd WP smoking session home visit, provide forms, urine cups package for week 2 of the study. WP Smoking Session 2. Days 1 through 7 are similar to session 1 with the exception that the RAs will add one tray of ice cubes and water in the WP jar. The RAs will arrange for a training session to use the charcoal-free electrically heated WP head. WP Smoking Session 3. Days 1 through 7 are similar to session 1 using room temperature water in the WP jar, however using the charcoal-free electrically heated WP head instead of using charcoal. During the last visit, the day after the 3rd smoking session, the RAs will interview participants to complete the Illnesses and Health Care History Form, pick up the final urine samples, and thank the participants.

ELIGIBILITY:
Inclusion Criteria for a Waterpipe Tobacco Smoker

* Adult male or female exclusive waterpipe tobacco smoker
* Smokes at least 1 waterpipe tobacco head per month
* Smokes waterpipe tobacco at home
* Age 21 years or older

Inclusion Criteria for a Non-Smoker

* Adult male or female non-smoker
* Lived in a 'non-smoker home' at least in the last month
* Age 21 years or older

Inclusion Criteria for a Non-Smoker Home

* No smokers have lived in in the past month
* No visitors had smoked indoors/outdoors in the past month

Exclusion Criteria

* Major physical/psychiatric illnesses
* Daily waterpipe smokers
* Pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nada Kassem, DrPH, Principal Investigator — San Diego State University
Locations (1):
- Center for Behavioral Epidemiology and Community Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kassem NO, Kassem NO, Liles S, Reilly E, Kas-Petrus F, Posis AIB, Hovell MF. Waterpipe device cleaning practices and disposal of waste associated with waterpipe tobacco smoking in homes in the USA. Tob Control. 2020 Feb;29(Suppl 2):s123-s130. doi: 10.1136/tobaccocontrol-2019-054959. Epub 2019 Jul 20. PMID 31326957

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We phone-screened 101 waterpipe tobacco (WPT) smoker respondents; 54 were eligible and were enrolled; 4 withdrew before the home visit (due to travel/change of mind).
  We phone-screened 51 non-smoker respondents; 31 were eligible and were enrolled; 1 non-smoker dropped out before the home visit (due to school/work schedule); 5 were excluded because of potential exposure to tobacco secondhand smoke (SHS) based on exhaled carbon monoxide (eCO) cut-off levels ≥3.6 ppm.(Deveci et al., 2004)
Groups:
- Waterpipe Tobacco (WPT) Smoking: In a repeated measures design, 50 adult male and female exclusive waterpipe tobacco (WPT) smokers will smoke weekly over a 3-week study period with 3 WPT smoking practices.
  WPT smoking: In a repeated measures design, 50 adult male and female exclusive WPT smokers will smoke WPT weekly over a 3-week study period with 3 WPT smoking practices as follows: 1) using room temperature water in the waterpipe (WP) jar, 2) adding ice cubes to the water in the WP jar, and 3) using a charcoal-free electronic WP head to heat the tobacco. Six Spot first morning urine samples will be provided by participants. Two urine samples per each of the 3 smoking sessions. Urine samples will be provided on the day of the WPT smoking session and the following day. Physiological measures will be taken at Baseline during the office visit and before and after each of the 3 WP tobacco smoking sessions.
- Control: A total of 25 adult male and female nonsmokers will be recruited as a control.
Period: Overall Study
Arm/Group | Waterpipe Tobacco (WPT) Smoking | Control
Started | 54 | 31
Completed | 50 | 25
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Protocol Violation | 0 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected only for retained participants (50 smokers; 25 non-smokers) in natural home settings (N=75), who were not disqualified or who were dropouts.
Groups:
- Waterpipe Smoking: 50 adult male and female exclusive waterpipe smokers will smoke waterpipe tobacco during a home smoking session
- Control: A total of 25 adult male and female nonsmokers will act as a control.
- Total: Total of all reporting groups
Arm/Group | Waterpipe Smoking | Control | Total
Number analyzed (Participants) | 54 | 31 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics were collected only for retained participants (50 smokers; 25 non-smokers) in natural home settings (N=75), who were not disqualified or who were dropouts.
  years
    number analyzed (Participants) | 50 | 25 | 75
    (all) | 25.3 (3.1) | 25.5 (4.6) | 25.3 (3.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics were collected only for retained participants (50 smokers; 25 non-smokers) in natural home settings (N=75), who were not disqualified or who were dropouts.
  Participants
    number analyzed (Participants) | 50 | 25 | 75
    Female | 25 | 13 | 38
    Male | 25 | 12 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics were collected only for retained participants (50 smokers; 25 non-smokers) in natural home settings (N=75), who were not disqualified or who were dropouts.
  Participants
    White, Caucasian, European: number analyzed (Participants) | 50 | 25 | 75
    White, Caucasian, European | 11 | 5 | 16
    Mexican, Hispanic, or Latino: number analyzed (Participants) | 50 | 25 | 75
    Mexican, Hispanic, or Latino | 16 | 8 | 24
    Black or African American: number analyzed (Participants) | 50 | 25 | 75
    Black or African American | 5 | 1 | 6
    Middle Eastern: number analyzed (Participants) | 50 | 25 | 75
    Middle Eastern | 13 | 0 | 13
    Asian/Multi-ethnic: number analyzed (Participants) | 50 | 25 | 75
    Asian/Multi-ethnic | 5 | 11 | 16
Highest level of education completed [Count of Participants; unit: Participants] — Population: Baseline characteristics were collected only for retained participants (50 smokers; 25 non-smokers) in natural home settings (N=75), who were not disqualified or who were dropouts.
  Participants
    High school: number analyzed (Participants) | 50 | 25 | 75
    High school | 7 | 1 | 8
    College, no degree: number analyzed (Participants) | 50 | 25 | 75
    College, no degree | 18 | 8 | 26
    College degree: number analyzed (Participants) | 50 | 25 | 75
    College degree | 25 | 15 | 40
    Missing: number analyzed (Participants) | 50 | 25 | 75
    Missing | 0 | 1 | 1
Type of natural home setting [Count of Participants; unit: Participants] — Population: Baseline characteristics were collected only for retained participants (50 smokers; 25 non-smokers) in natural home settings (N=75), who were not disqualified or who were dropouts.
  Participants
    House: number analyzed (Participants) | 50 | 25 | 75
    House | 30 | 12 | 42
    Apartment/Townhouse: number analyzed (Participants) | 50 | 25 | 75
    Apartment/Townhouse | 19 | 13 | 32
    Missing Data: number analyzed (Participants) | 50 | 25 | 75
    Missing Data | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparing Cotinine Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: Investigators will assess change in creatinine-adjusted urinary levels of cotinine (a metabolite of the addictive drug nicotine) in ng/mL, from pre-to post, at each of 2 waterpipe tobacco smoking sessions. For each of the 2 smoking sessions, smokers will provide two first morning spot urine samples--the day of the smoking session and the following morning. The two waterpipe tobacco smoking sessions are as follows: 1) using charcoal to heat the tobacco, and 2) using a charcoal-free electronic waterpipe head to heat the tobacco.
Time Frame: On 2 days for each of two smoking sessions, smokers will provide 2 first morning spot urine samples--one urine sample on the morning of the day of the smoking session, and one urine sample on the morning of the following day.
Population: Participants will be recruited via intercept interviews from San Diego County, CA communities. Inclusion Criteria for Participants: 1) Adult waterpipe smoker: A male or female, 18 years or older, who smokes WP tobacco exclusively, smokes at least 1 WP head per month, and smokes at least 1 WP head per WP smoking session, smokes WP at home, agrees to smoke Starbuzz WP tobacco, and lives in a 'smoker home'; 2) Adult non-smoker: A male or female, 18 years or older, who lives in a 'non-smoker home'.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Charcoal-heated Waterpipe Smoking; Electric-head-heated Waterpipe Smoking: In a repeated measures design, 50 adult male and female exclusive WP smokers will smoke WP tobacco during the smoking session at their own home, using the traditional charcoal to heat the tobacco.
  Two spot first morning urine samples will be provided by participants. Urine samples will be provided on the day of the WP tobacco smoking session and on the following day. Physiological measures will be taken before and after the WP tobacco smoking session.
Arm/Group | Charcoal-heated Waterpipe Smoking | Electric-head-heated Waterpipe Smoking
Number analyzed (Participants) | 50 | 50
ng/mL | 34.9 [24.2 to 50.5] | 26.4 [18.3 to 38.0]
Statistical Analysis 1: Comparison: Charcoal-heated Waterpipe Smoking vs Electric-head-heated Waterpipe Smoking; Test type: Other; p = 0.115, Wilcoxon signed-rank test; z score = 1.578; We used the Wilcoxon signed-rank test (two-tailed alpha level p < 0.05), appropriate for within-subjects tests, to determine whether the pre-to-post change in biomarker levels for the Charcoal-heated tobacco smoking session (n=50) significantly different from the pre-to-post change in biomarker levels for the Electric Head-heated tobacco smoking session (using the same 50 participants after a weeklong washout period)

2. Primary Outcome: Comparing S-phenyl-mercapturic Acid (SPMA) Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: Investigators will assess change in creatinine-adjusted urinary levels of SPMA (a metabolite of the human hematotoxicant and leukemogen benzene) in pmol/mL, from pre-to post, at each of 2 waterpipe tobacco smoking sessions. For each of the 2 smoking sessions, smokers will provide two first morning spot urine samples--the day of the smoking session and the following morning. The two waterpipe tobacco smoking sessions are as follows: 1) using charcoal to heat the tobacco, and 2) using a charcoal-free electronic waterpipe head to heat the tobacco.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Charcoal-heated Waterpipe Smoking | Electric-head-heated Waterpipe Smoking
Number analyzed (Participants) | 50 | 50
pmol/mL | 1.35 [0.78 to 2.30] | 0.34 [0.20 to 0.57]
Statistical Analysis 1: Comparison: Charcoal-heated Waterpipe Smoking vs Electric-head-heated Waterpipe Smoking; Test type: Other; p = 0.619, z; z = 0.497; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Comparing 1-hydroxypyrene (1-HOP) But Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: Investigators will assess change in creatinine-adjusted urinary levels of 1-HOP (a metabolite of the genotoxic carcinogen pyrene) in pmol/ML, from pre-to post, at each of 2 waterpipe tobacco smoking sessions. For each of the 2 smoking sessions, smokers will provide two first morning spot urine samples--the day of the smoking session and the following morning. The two waterpipe tobacco smoking sessions are as follows: 1) using charcoal to heat the tobacco, and 2) using a charcoal-free electronic waterpipe head to heat the tobacco.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ML
Arm/Group | Charcoal-heated Waterpipe Smoking | Electric-head-heated Waterpipe Smoking
Number analyzed (Participants) | 50 | 50
pmol/ML | 0.47 [0.34 to 0.65] | 0.48 [0.35 to 0.66]
Statistical Analysis 1: Comparison: Charcoal-heated Waterpipe Smoking vs Electric-head-heated Waterpipe Smoking; Test type: Other; p = 0.085, Wilcox and signed rank test; z = 1.720; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Comparing Exhaled Carbon Monoxide Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: measuring exhaled CO using a Micro+ Smokerlyzer® carbon monoxide (CO) monitor for exhaled CO before and after each of two waterpipe tobacco smoking sessions, investigators will determine the differential change, pre-to-post waterpipe tobacco smoking, between heating by charcoal vs heating by electric head
Time Frame: Assessment will be taken immediately before starting to smoke, and immediately at conclusion of each of the 2 smoking sessions.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Parts per million
Arm/Group | Charcoal-heated Waterpipe Smoking | Electric-head-heated Waterpipe Smoking
Number analyzed (Participants) | 50 | 50
Parts per million | 107 [84 to 136] | 3.5 [2.5 to 4.9]
Statistical Analysis 1: Comparison: Charcoal-heated Waterpipe Smoking vs Electric-head-heated Waterpipe Smoking; Test type: Other; p < 0.001, Wilcoxon signed rank test; z = 6.154; [other analysis details as in outcome 1, analysis 1]

5. Primary Outcome: Comparing Systolic Blood Pressure Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: The investigators will determine the differential effects of WP smoking practices on change in systolic blood pressure in mm/Hg after each of two WP smoking sessions: 1) using charcoal to heat the tobacco, and 2) using a charcoal-free electronic waterpipe head to heat the tobacco.
Time Frame: Systolic & diastolic blood pressure and heart rate were assessed multiple times (at intervals>1 min) and averaged. Assessments were at the start and end of each smoking session (mean duration=31 min).
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mmHg (Millimeters of mercury)
Groups:
- Waterpipe Smoking - Charcoal: In a repeated measures design, 50 adult male and female exclusive WP smokers will smoke WP tobacco weekly over a 3-week study period with 3 WP smoking practices.
  Waterpipe smoking: In a repeated measures design, 50 adult male and female exclusive WP tobacco smokers will smoke WP tobacco weekly over a 3-week study period with 3 WP smoking practices as follows: 1) using room temperature water in the WP jar, 2) adding ice cubes to the water in the WP jar, and 3) using a charcoal-free electronic WP head to heat the tobacco. Six Spot first morning urine samples will be provided by participants. Two urine samples per each of the 3 smoking sessions. Urine samples will be provided on the day of the WP tobacco smoking session and the following day. Physiological measures will be taken at Baseline during the office visit and before and after each of the 3 WP tobacco smoking sessions.
- Waterpipe Smoking - Electric Head: In a repeated measures design, 50 adult male and female exclusive WP smokers will smoke WP tobacco weekly over a 3-week study period with 3 WP smoking practices.
  Waterpipe smoking: In a repeated measures design, 50 adult male and female exclusive WP tobacco smokers will smoke WP tobacco weekly over a 2-week study period with 2 WP smoking practices as follows: 1) using charcoal to heat the tobacco, 2) using a charcoal-free electronic WP head to heat the tobacco. Physiological measures will be taken before and after each of the 2 WP tobacco smoking sessions.
Arm/Group | Waterpipe Smoking - Charcoal | Waterpipe Smoking - Electric Head
Number analyzed (Participants) | 50 | 50
mmHg (Millimeters of mercury) | 122 [118 to 125] | 120 [116 to 124]
Statistical Analysis 1: Comparison: Waterpipe Smoking - Charcoal vs Waterpipe Smoking - Electric Head; Test type: Other; p = 0.253, Wilcoxon signed rank test; z = -1.144; We used the Wilcoxon signed-rank test (two-tailed alpha level p < 0.05), appropriate for within-subjects tests, to determine whether the pre-to-post change in systolic blood pressure for the Charcoal-heated tobacco smoking session (n=50) significantly different from the pre-to-post change in biomarker levels for the Electric Head-heated tobacco smoking session (using the same 50 participants after a weeklong washout period)

6. Primary Outcome: Comparing Diastolic Blood Pressure Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: The investigators will investigate the differential effects of WP smoking practices on change in diastolic blood pressure in mm/Hg after each of two WP smoking sessions: 1) using charcoal to heat the tobacco, and 2) using a charcoal-free electronic waterpipe head to heat the tobacco.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mmHg (Millimeters of mercury)
Groups:
- Charcoal-heated Waterpipe Smoking; Electric-head-heated Waterpipe Smoking: In a repeated measures design, 50 adult male and female exclusive WP smokers will smoke WP tobacco during the smoking session at their own home, using the traditional charcoal to heat the tobacco.
Arm/Group | Charcoal-heated Waterpipe Smoking | Electric-head-heated Waterpipe Smoking
Number analyzed (Participants) | 50 | 50
mmHg (Millimeters of mercury) | 79 [77 to 81] | 78 [76 to 80]
Statistical Analysis 1: Comparison: Charcoal-heated Waterpipe Smoking vs Electric-head-heated Waterpipe Smoking; Test type: Other; p = 0.315, Wilcoxon signed rank test; z = -1.004; We used the Wilcoxon signed-rank test (two-tailed alpha level p < 0.05), appropriate for within-subjects tests, to determine whether the pre-to-post change in diastolic blood pressure for the Charcoal-heated tobacco smoking session (n=50) significantly different from the pre-to-post change in diastolic blood pressure for the Electric Head-heated tobacco smoking session (using the same 50 participants after a weeklong washout period)

7. Primary Outcome: Comparing Heart Rate Pre-to-post Change Between 2 Waterpipe Smoking Sessions: Heating Waterpipe Tobacco by (a) Charcoal vs (b) an Electric Head
Description: The investigators will investigate the differential effects of WP smoking practices on change in heart rate in beats per minute after each of two WP smoking sessions: 1) using charcoal to heat the tobacco, and 2) using a charcoal-free electronic waterpipe head to heat the tobacco.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Heart beats/minute
Arm/Group | Charcoal-heated Waterpipe Smoking | Electric-head-heated Waterpipe Smoking
Number analyzed (Participants) | 50 | 50
Heart beats/minute | 80 [76 to 83] | 77 [73 to 80]
Statistical Analysis 1: Comparison: Charcoal-heated Waterpipe Smoking vs Electric-head-heated Waterpipe Smoking; Test type: Other; p = 0.002, Wilcox and signed rank test; z = 3.089; We used the Wilcoxon signed-rank test (two-tailed alpha level p < 0.05), appropriate for within-subjects tests, to determine whether the pre-to-post change in heart rate for the Charcoal-heated tobacco smoking session (n=50) was significantly different from the pre-to-post change in heart rate for the Electric Head-heated tobacco smoking session (using the same 50 participants after a weeklong washout period)

8. Primary Outcome: Assess Difference in Cotinine Levels Between (a) Non-smokers vs. (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: Investigators will assess change in creatinine-adjusted urinary levels of cotinine (a metabolite of nicotine) in ng/mL, For a smoking session using charcoal to heat the tobacco, waterpipe smokers will provide two first morning spot urine samples--the morning of the day of the smoking session and the morning of the following day. The investigators will assess difference in urinary cotinine levels between (a) non-smokers vs. (b) waterpipe tobacco smokers after the waterpipe smoking session.
Time Frame: For smokers: Early morning on the smoking session day to early morning the day after. For non-smokers: early in the morning of the home visit.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Waterpipe Smoking - Charcoal Heated: 50 adult male and female exclusive waterpipe smokers will smoke waterpipe tobacco during a home smoking session
- Control: A total of 25 adult male and female nonsmokers were recruited as a control.
Arm/Group | Waterpipe Smoking - Charcoal Heated | Control
Number analyzed (Participants) | 50 | 25
ng/mL | 34.9 [24.2 to 50.5] | 0.02 [0.01 to 0.04]
Statistical Analysis 1: Comparison: Waterpipe Smoking - Charcoal Heated vs Control; Test type: Other; p < 0.001, Mann-Whitney U rank sum test; z = -7.024; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of the cotinine metabolite after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

9. Primary Outcome: Assess Difference in SPMA Levels Between (a) Non-smokers and (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: Investigators will assess change in creatinine-adjusted levels of SPMA (a metabolite of the human hematotoxicant and leukemogen benzene) in pmol/mL, For a smoking session using charcoal to heat the tobacco, waterpipe smokers will provide two first morning spot urine samples--the morning of the day of the smoking session and the morning of the following day. The investigators will assess difference in urinary cotinine levels between (a) non-smokers vs. (b) waterpipe tobacco smokers after the waterpipe smoking session.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/mL | 1.35 [0.78 to 2.30] | 0.17 [0.11 to 0.27]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p < 0.001, Mann-Whitney U rank sum test; z = -4.541; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of the SPMA metabolite after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

10. Primary Outcome: Assess Difference in 1-HOP Levels Between (a) Non-smokers and (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: Investigators will assess change in creatinine-adjusted urinary levels of 1-HOP (metabolite of the genotoxic carcinogen pyrene in pmol/mL, For a smoking session using charcoal to heat the tobacco, waterpipe smokers will provide two first morning spot urine samples--the morning of the day of the smoking session and the morning of the following day. The investigators will assess difference in urinary cotinine levels between (a) non-smokers vs. (b) waterpipe tobacco smokers after the waterpipe smoking session.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/mL | 0.47 [0.34 to 0.65] | 0.23 [0.16 to 0.35]
Statistical Analysis 1: Comparison: Waterpipe Smoking; Test type: Other; p = .010, Mann-Whitney U rank sum test; z = -2.569; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of the 1-HOP metabolite after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

11. Primary Outcome: Assess Difference in Exhaled Carbon Monoxide Levels Between (a) Non-smokers and (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: measuring exhaled CO using a Micro+ Smokerlyzer® CO monitor for exhaled CO before and after the heating by charcoal waterpipe tobacco smoking session, investigators will compare the levels between (a) non-smokers and (b) waterpipe tobacco smokers after their smoking session
Time Frame: For the smokers: Assessment will be taken immediately before starting to smoke, and immediately at conclusion of each of the smoking session. For the non-smokers: Assessment will be taken at the home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Parts per million
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
Parts per million | 107 [84 to 136] | 2.8 [2.1 to 3.6]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p < 0.001, Mann-Whitney U rank sum test; z = -7.030; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of the exhaled carbon monoxide after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

12. Primary Outcome: Assess Difference in Systolic Blood Pressure Levels Between (a) Non-smokers and (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: measuring systolic blood pressure levels before and after the waterpipe tobacco smoking session, investigators will compare the levels between (a) non-smokers and (b) waterpipe tobacco smokers after their smoking session
Time Frame: Systolic & diastolic blood pressure and heart rate were assessed multiple times (at intervals>1 min) and averaged. Assessments were at the start and end of each smoking session (mean duration =31 min), or at one point during the non-smoker home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Millimeters of mercury
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
Millimeters of mercury | 122 [118 to 125] | 117 [111 to 124]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.192, Mann-Whitney U test; z = -1.304; [other analysis details as in outcome 8, analysis 1]

13. Primary Outcome: Assess Difference in Diastolic Blood Pressure Levels Between (a) Non-smokers and (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: measuring diastolic blood pressure levels before and after the waterpipe tobacco smoking session, investigators will compare the levels between (a) non-smokers and (b) waterpipe tobacco smokers after their smoking session
Time Frame: as for outcome 12
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Millimeters of mercury
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
Millimeters of mercury | 79 [77 to 81] | 75 [73 to 78]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.033, Mann-Whitney U rank sum test; z = -2.136; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level diastolic blood pressure after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

14. Primary Outcome: Assess Difference in Heart Rate Levels Between (a) Non-smokers and (b) Smokers Post a Waterpipe Smoking Session, Using Tobacco Heated by Charcoal
Description: measuring heart rate levels before and after the waterpipe tobacco smoking session, investigators will compare the levels between (a) non-smokers and (b) waterpipe tobacco smokers after their smoking session
Time Frame: as for outcome 12
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
Beats per minute | 80 [76 to 83] | 76 [71 to 81]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.223, Mann-Whitney U rank sum test; z = -1.220; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of the heart rate after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

15. Primary Outcome: Assess Difference in Cotinine Levels Between (a) Non-smokers vs. (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: Investigators will assess creatinine-adjusted urinary levels of cotinine (a metabolite of nicotine) in ng/mL.
  For a smoking session using an electric head to heat the tobacco, waterpipe smokers will provide two first morning spot urine samples--the morning of the day of the smoking session and the morning of the following day. The investigators will compare (a) non-smoker levels with (b) waterpipe tobacco smoker levels after their waterpipe smoking session.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (99% Confidence Interval); unit: ng/mL
Groups:
- Control: 25 adult male and female nonsmokers will act as a control
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
ng/mL | 26.4 [18.3 to 38] | 0.02 [0.01 to 0.04]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p < 0.001, Mann Whitney U rank sum test; z = -7.024; [other analysis details as in outcome 8, analysis 1]

16. Primary Outcome: Assess Difference in SPMA Levels Between (a) Non-smokers and (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: Investigators will assess creatinine-adjusted urinary levels of SPMA (a metabolite of benzene) in pmol/mL.
  For a smoking session using an electric head to heat the tobacco, waterpipe smokers will provide two first morning spot urine samples--the morning of the day of the smoking session and the morning of the following day. The investigators will compare (a) non-smoker levels with (b) waterpipe tobacco smoker levels after their waterpipe smoking session.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/mL | 0.34 [0.20 to 0.57] | 0.17 [0.11 to 0.27]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.212, Mann-Whitney U rank sum test; z = -1.248; [other analysis details as in outcome 9, analysis 1]

17. Primary Outcome: Assess Difference in 1-HOP Levels Between (a) Non-smokers and (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: Investigators will assess creatinine-adjusted urinary levels of 1-HOP (a metabolite of pyrene, a polycyclic aromatic hydrocarbon) pmol/ML.
  For a smoking session using an electric head to heat the tobacco, waterpipe smokers will provide two first morning spot urine samples--the morning of the day of the smoking session and the morning of the following day. The investigators will compare (a) non-smoker levels with (b) waterpipe tobacco smoker levels after their waterpipe smoking session.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/mL | 0.48 [0.35 to 0.66] | 0.23 [0.16 to 0.35]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.007, Mann-Whitney U rank sum test; z = -2.721; [other analysis details as in outcome 8, analysis 1]

18. Primary Outcome: Assess Difference in Exhaled Carbon Monoxide Levels Between (a) Non-smokers and (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: measuring exhaled carbon monoxide levels before and after the waterpipe tobacco smoking session, investigators will compare the levels between (a) non-smokers and (b) waterpipe tobacco smokers after their smoking session
Time Frame: For the smokers: Assessment will be taken immediately before starting to smoke, and immediately at conclusion of the smoking session. For the non-smokers: Assessment will be taken at the home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Parts per million
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
Parts per million | 3.5 [2.5 to 4.9] | 2.8 [2.1 to 3.6]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.006, Mann-Whitney U rank sum test; z = 2.778; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of exhaled carbon monoxide after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

19. Primary Outcome: Assess Difference in Systolic Blood Pressure Levels Between (a) Non-smokers and (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: For a smoking session using an electric head to heat the tobacco, investigators will measure systolic blood pressure levels before and after the waterpipe tobacco smoking session, and compare (a) non-smoker levels with (b) waterpipe tobacco smoker levels after their waterpipe smoking session.
Time Frame: as for outcome 12
Population: Waterpipe smoking: 50 adult male and female exclusive waterpipe smokers will smoke waterpipe tobacco during a home smoking session Control: A total of 25 adult male and female nonsmokers were recruited as a control.
Measure: Geometric Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
mmHg | 120 [116 to 124] | 117 [111 to 124]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.406, Mann-Whitney U rank sum test; z = -0.832; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of systolic blood pressure after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

20. Primary Outcome: Assess Difference in Diastolic Blood Pressure Levels Between (a) Non-smokers and (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: For a smoking session using an electric head to heat the tobacco, investigators will measure diastolic blood pressure levels before and after the waterpipe tobacco smoking session, and compare (a) non-smoker levels with (b) waterpipe tobacco smoker levels after their waterpipe smoking session.
Time Frame: Systolic & diastolic blood pressure and heart rate were assessed multiple times (at intervals>1 min) and averaged. Assessments were at the start and end of each smoking session (mean duration=31 min), or at one point during the non-smoker home visit.
Measure: Geometric Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
mmHg | 78 [76 to 80] | 75 [73 to 78]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.142, Mann-Whitney U ranksum test; z = -1.467; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of diastolic blood pressure after a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

21. Primary Outcome: Assess Difference in Heart Rate Levels Between (a) Non-smokers and (b) Smokers After a Waterpipe Smoking Session, Using Tobacco Heated by an Electric Head
Description: For a smoking session using an electric head to heat the tobacco, investigators will measure heart rate levels before and after the waterpipe tobacco smoking session, and compare (a) non-smoker levels with (b) waterpipe tobacco smoker levels after their waterpipe smoking session.
Time Frame: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
Beats per minute | 77 [73 to 80] | 76 [71 to 81]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.551, Mann-Whitney U rank sum test; z = -0.596; [other analysis details as in outcome 14, analysis 1]

22. Secondary Outcome: Assess Difference in Urinary L-2-(Acetylamino)-6-(2,5-dihydro-2-oxo-1H-pyrrol-1-yl)-1-hexanoic Acid (Furan-BDA-NAL) Between Levels at Post Waterpipe Tobacco Smoking Versus Non-smoker Levels.
Description: The investigators will assess difference in urinary Furan-BDA-NAL levels between non-smokers and post a smoking session for waterpipe tobacco smokers. Furan-BDA-NAL is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples: for smokers, the day of the smoking session and the day following the smoking session; for non-smokers, the day of the home visit.
Time Frame: For smokers: Early morning on day 1 to early morning on day 2. For non-smokers: early in the morning of the home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ML
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/ML | 131 [111 to 155] | 112 [91 to 139]
Statistical Analysis 1: Comparison: Waterpipe Smoking; Test type: Other; p = 0.431, Mann-Whitney U rank sum test; z = -0.787; We used the Mann-Whitney U rank sum test (two-tailed alpha level p < 0.05), appropriate for between-subjects analyses, to determine whether level of the furan metabolite post a tobacco smoking session for n=50 smokers differed from the level for n=25 non-smokers

23. Secondary Outcome: Assess Difference in Urinary Furan-BDA-Lys Between Levels at Post Waterpipe Tobacco Smoking Versus Non-smoker Levels.
Description: The investigators will assess difference in urinary Furan-BDA-Lys levels between non-smokers and post a smoking session for waterpipe tobacco smokers. Furan-BDA-Lysis a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples: for smokers, the day of the smoking session and the day following the smoking session; for non-smokers, the day of the home visit.
Time Frame: For smokers: Early morning on day 1 to early morning on day 2. For non-smokers: early in the morning of the home visit.
Population: Participants will be recruited via intercept interviews from San Diego County, CA communities. Inclusion Criteria for Participants: A adult male or female, 18 years or older, who smokes WP tobacco exclusively, smokes at least 1 WP head per month, and smokes at least 1 WP head per WP smoking session, smokes WP at home, agrees to smoke Starbuzz WP tobacco, and lives in a 'smoker home'
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ML
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/ML | 47 [36 to 60] | 44 [34 to 57]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.515, Mann-Whitney U rank sum test; z = -0.652; [other analysis details as in outcome 22, analysis 1]

24. Secondary Outcome: Assess Difference in Urinary N-acetyl-S-[1-(5-acetylamino-5-carboxylpentyl)-1H-pyrrol-3-yl]-L-cysteine (Furan-NAC-BDA-NAL) Between Levels at Post Waterpipe Tobacco Smoking Versus Non-smoker Levels.
Description: The investigators will assess difference in urinary Furan-NAC-BDA-NAL levels between non-smokers and post a smoking session for waterpipe tobacco smokers. Furan-NAC-BDA-NAL is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples: for smokers, the day of the smoking session and the day following the smoking session; for non-smokers, the day of the home visit.
Time Frame: For smokers: Early morning on day 1 to early morning on day 2. For non-smokers: early in the morning of the home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ML
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/ML | 0.05 [0.04 to 0.07] | 0.01 [0.00 to 0.03]
Statistical Analysis 1: Comparison: Waterpipe Smoking; Test type: Other; p = 0. 017, Mann-Whitney U rank sum test; z = -2.394; [other analysis details as in outcome 22, analysis 1]

25. Secondary Outcome: Assess Difference in Urinary N-acetyl-S-[1-(5-amino-5-carboxylpentyl)-1H-pyrrol-3-yl]-L-cysteine (Furan-NAC-BDA-Lys) Between Levels at Post Waterpipe Tobacco Smoking Versus Non-smoker Levels.
Description: The investigators will assess difference in urinary Furan-NAC-BDA-Lys levels between non-smokers and post a smoking session for waterpipe tobacco smokers. Furan-BNAC-BDA-Lys is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples: for smokers, the day of the smoking session and the day following the smoking session; for non-smokers, the day of the home visit.
Time Frame: For smokers: Early morning on day 1 to early morning on day 2. For non-smokers: early in the morning of the home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/mL | 4.0 [3.5 to 4.6] | 2.4 [1.1 to 5.3]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.199, Mann-Whitney U rank sum test; z = -1.286; [other analysis details as in outcome 22, analysis 1]

26. Secondary Outcome: Assess Difference in Urinary Furan-NAC-BDA-Lys Sulfoxide' Between Levels at Post Waterpipe Tobacco Smoking Versus Non-smoker Levels.
Description: The investigators will assess difference in urinary Furan-NAC-BDA-Lys sulfoxide levels between non-smokers and post a smoking session for waterpipe tobacco smokers. Furan-NAC-BDA-Lys sulfoxide is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples: for smokers, the day of the smoking session and the day following the smoking session; for non-smokers, the day of the home visit.
Time Frame: For smokers: Early morning on day 1 to early morning on day 2. For non-smokers: early in the morning of the home visit.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ML
Arm/Group | Waterpipe Smoking | Control
Number analyzed (Participants) | 50 | 25
pmol/ML | 3.1 [2.6 to 3.6] | 2.1 [1.8 to 2.5]
Statistical Analysis 1: Comparison: Waterpipe Smoking vs Control; Test type: Other; p = 0.002, Mann-Whitney U rank sum test; z = -3.091; [other analysis details as in outcome 22, analysis 1]

27. Secondary Outcome: Assess Difference in Urinary Furan-BDA-NAL Between Levels Pre the Waterpipe Tobacco Smoking Session vs Post the Waterpipe Tobacco Smoking Session.
Description: Investigators will assess difference between pre-smoking session levels of urinary Furan-BDA-NAL in waterpipe tobacco smokers and post that smoking session. Furan-BDA-NAL is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples, the day of the smoking session and the day following the smoking session.
Time Frame: Early morning on day 1 to early morning on day 2.
Population: Participants were recruited via intercept interviews from San Diego County, CA communities. Inclusion Criteria for Participants: A male or female adult waterpipe smoker, 18 years or older, who smokes WP tobacco exclusively, smokes at least 1 WP head per month, and smokes at least 1 WP head per WP smoking session, smokes WP at home, agrees to smoke Starbuzz WP tobacco, and lives in a 'smoker home'.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Groups:
- Waterpipe Smokers, Pre the Smoking Session: Pre-session: 50 adult male and female exclusive waterpipe smokers, who will provide a first morning spot urine sample prior to a home smoking session
- Waterpipe Smokers, Post the Smoking Session: Post-session: The same 50 adult male and female exclusive waterpipe smokers will also provide a first morning spot urine sample on the morning after the home smoking session
Arm/Group | Waterpipe Smokers, Pre the Smoking Session | Waterpipe Smokers, Post the Smoking Session
Number analyzed (Participants) | 50 | 50
pmol/mL | 128 [111 to 148] | 131 [111 to 155]
Statistical Analysis 1: Comparison: Waterpipe Smokers, Pre the Smoking Session vs Waterpipe Smokers, Post the Smoking Session; Test type: Other; p = 0.896, Wilcoxon signed rank test; z = 0.130; We used the Wilcoxon signed rank test (two-tailed alpha level p < 0.05), appropriate for within-subjects analyses, to determine whether level of the furan metabolite post a tobacco smoking session for n=50 smokers differed from the level pre the tobacco smoking session

28. Secondary Outcome: Assess Difference in Urinary Furan-BDA-Lys Between Levels Pre the Waterpipe Tobacco Smoking Session vs Post the Waterpipe Tobacco Smoking Session.
Description: Investigators will assess difference between pre-smoking session levels of urinary Furan-BDA-Lys in waterpipe tobacco smokers and post that smoking session. Furan-BDA-Lys is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples, the day of the smoking session and the day following the smoking session.
Time Frame: Early morning on day 1 to early morning on day 2
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smokers, Pre the Smoking Session | Waterpipe Smokers, Post the Smoking Session
Number analyzed (Participants) | 50 | 50
pmol/mL | 42 [32 to 55] | 47 [36 to 60]
Statistical Analysis 1: Comparison: Waterpipe Smokers, Pre the Smoking Session vs Waterpipe Smokers, Post the Smoking Session; Test type: Other; p = 0.717, The Wilcoxon signed rank test; z = -0.362; [other analysis details as in outcome 27, analysis 1]

29. Secondary Outcome: Assess Difference in Urinary Furan-NAC-BDA-NAL Between Levels Pre the Waterpipe Tobacco Smoking Session vs Post the Waterpipe Tobacco Smoking Session
Description: Investigators will assess difference between pre-smoking session levels of urinary Furan-NAC-BDA-NAL in waterpipe tobacco smokers and post that smoking session. Furan-NAC-BDA-NAL is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples, the day of the smoking session and the day following the smoking session.
Time Frame: Early morning on day 1 to early morning on day 2
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smokers, Pre the Smoking Session | Waterpipe Smokers, Post the Smoking Session
Number analyzed (Participants) | 50 | 50
pmol/mL | 0.06 [0.04 to 0.09] | 0.05 [0.04 to 0.07]
Statistical Analysis 1: Comparison: Waterpipe Smokers, Pre the Smoking Session vs Waterpipe Smokers, Post the Smoking Session; Test type: Other; p = 0.026, Wilcoxon signed rank test; z = 2.233; [other analysis details as in outcome 27, analysis 1]

30. Secondary Outcome: Assess Difference in Urinary Furan-NAC-BDA-Lys Between Levels Pre the Waterpipe Tobacco Smoking Session vs Post the Waterpipe Tobacco Smoking Session
Description: Investigators will assess difference between pre-smoking session levels of urinary Furan-NAC-BDA-Lys in waterpipe tobacco smokers and post that smoking session. Furan-NAC-BDA-Lys is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples, the day of the smoking session and the day following the smoking session.
Time Frame: Early morning on day 1 to early morning on day 2
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smokers, Pre the Smoking Session | Waterpipe Smokers, Post the Smoking Session
Number analyzed (Participants) | 50 | 50
pmol/mL | 4.0 [3.5 to 4.6] | 4.0 [3.5 to 4.6]
Statistical Analysis 1: Comparison: Waterpipe Smokers, Pre the Smoking Session vs Waterpipe Smokers, Post the Smoking Session; Test type: Other; p = 0.702, Wilcoxon signed rank test; z = 0.383; [other analysis details as in outcome 27, analysis 1]

31. Secondary Outcome: Assess Difference in Urinary Furan-NAC-BDA-Lys Sulfoxide Between Levels Pre the Waterpipe Tobacco Smoking Session vs Post the Waterpipe Tobacco Smoking Session
Description: Investigators will assess difference between pre-smoking session levels of urinary Furan-NAC-BDA-Lys sulfoxide in waterpipe tobacco smokers and post that smoking session. Furan-NAC-BDA-Lys sulfoxide is a metabolite of furan, a liver toxicant and carcinogen. It will be collected for laboratory assay using two first morning spot urine samples, the day of the smoking session and the day following the smoking session
Time Frame: Early morning on day 1 to early morning on day 2
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/mL
Arm/Group | Waterpipe Smokers, Pre the Smoking Session | Waterpipe Smokers, Post the Smoking Session
Number analyzed (Participants) | 50 | 50
pmol/mL | 3.4 [2.9 to 4.1] | 3.1 [2.6 to 3.6]
Statistical Analysis 1: Comparison: Waterpipe Smokers, Pre the Smoking Session vs Waterpipe Smokers, Post the Smoking Session; Test type: Other; p = 0.025, Wilcoxon signed rank test; z = 2.244; [other analysis details as in outcome 27, analysis 1]

ADVERSE EVENTS:
Time Frame: For each of the 50 participants sequentially enrolled as a hookah smoker, the duration of their participation in the study, from enrollment to exit, was three weeks. For each of the 25 participants sequentially enrolled as a non-smoker, the duration of their participation in the study, from enrollment to exit, was one week.
Arm/Group | Waterpipe Smoking | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 0/50 | 0/25

LIMITATIONS AND CAVEATS:
Smoking duration was shorter for electric head vs charcoal, reducing smoke exposure. WPT smokers smoked alone, not socially, generating less sidestream smoke exposure. Spot urine samples may have underestimated peak levels of benzene and pyrene, due to half-lifes differing among metabolites. Participant use of one type of charcoal, tobacco, WP hoses, and electric heater; convenience sampling; n=50; and participant age 21-35, suggest data may not be representative of WPT smokers in general.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03253653/Prot_SAP_ICF_001.pdf